CLINICAL TRIAL: NCT06177119
Title: Timing of Administration of Systemic Antibiotics Associated With Scaling and Root Planing in the Treatment of Periodontitis: Clinical and Microbiological Evaluation
Brief Title: Amoxicillin and Metronidazole During or After the Periodontal Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Belén Retamal-Valdes (Other)
Responsible Party: Sponsor-Investigator, Belén Retamal-Valdes, Professor, University of Guarulhos
Organization: University of Guarulhos (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SISNEP/726_Jan31_2012
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Periodontitis
Keywords: periodontitis; scaling and root planing; metronidazole; amoxicillin; treatment; microbiota
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test 1 (Experimental): Scaling and root planing + Metronidazole (400 mg/thrice a day,TID) and Amoxicillin (500 mg/ TID) for 14 days, starting with the first SRP session
  Interventions: Procedure: Scaling and root planing; Drug: Placebos after SRP; Drug: Metronidazole during SRP; Drug: Amoxicillin during SRP
- Test 2 (Experimental): Scaling and root planing (SRP) + Metronidazole (400 mg/thrice a day,TID) and Amoxicillin (500 mg/ TID) immediately after the end of the SRP in the following 14 days.
  Interventions: Procedure: Scaling and root planing; Drug: Placebos during SRP; Drug: Metronidazole after SRP; Drug: Amoxicillin after SRP

INTERVENTIONS:
Procedure: Scaling and root planing — SRP will be performed in four to six appointments lasting approximately 1 h each, using manual curettes (Hu-Friedy, Chicago, IL, USA) and ultrasonic device (Cavitron Select SPC, Dentsply professional, York, PA, USA) under local anesthesia. The deep sites will be scaled throughout the first week and treatment of the entire oral cavity will be completed in 14 days.
  Other Names: SRP
Drug: Placebos during SRP — Amoxicillin and metronidazole placebos thrice a day for 14 days, beginning with the first SRP session.
  Arms: Test 2
Drug: Placebos after SRP — Amoxicillin and metronidazole placebos thrice a day for 14 days, beginning after the last SRP session.
  Arms: Test 1
Drug: Metronidazole during SRP — Metronidazole 400 mg, thrice a day for 14 days, beginning with the first SRP session.
  Arms: Test 1
Drug: Amoxicillin during SRP — Amoxicillin 500 mg, thrice a day for 14 days, beginning with the first SRP session.
  Arms: Test 1
Drug: Metronidazole after SRP — Metronidazole 400 mg, thrice a day for 14 days, beginning after the last SRP session.
  Arms: Test 2
Drug: Amoxicillin after SRP — Amoxicillin 500 mg, thrice a day for 14 days, beginning after the last SRP session.
  Arms: Test 2

SUMMARY:
This randomized clinical trial aimed to compare the clinical and microbiological effects of different times of administration of metronidazole (MTZ) and amoxicillin (AMX) in the treatment of periodontitis.

DETAILED DESCRIPTION:
Scaling and root planing (SRP) is the most used periodontal therapy for periodontal treatment. Despite leading, in most cases, to an improvement in periodontal clinical parameters, SRP is often insufficient to profoundly modify the pathogenic bacterial profile to a profile related to periodontal health, especially in cases of more advanced and generalized diseases. Thus, other therapies supporting SRP, such as systemic antibiotics, have been proposed with the aim of enhancing the clinical and microbiological effects of this form of therapy. Studies have shown excellent clinical and microbiological results using the association of systemic antibiotics, especially the association of metronidazole (MTZ) and amoxicillin (AMX) in the treatment of severe periodontitis. However, some essential issues associated with the use of these antibiotics remain to be established. Therefore, the aim of this randomized clinical trial was to compare the clinical and microbiological effects of different times of administration of metronidazole (MTZ) and amoxicillin (AMX) in the treatment of periodontitis. Seventy-two subjects with severe periodontitis were selected and randomized into two groups (n = 36 / group) - Test 1 (T1): SRP in 14 days, associated with the concomitant use of AMX (500mg, 3x / day) and MTZ (400mg 3x / day) for 14 days; and Test 2 (T2): SRP in 14 days, associated with the use of AMX and MTZ immediately after the end of the SRP in the following 14 days. All volunteers received clinical and microbiological evaluation at baseline, 3, 6 and 12 months post-SRP. Subgingival biofilm samples were collected by subject and analyzed for counts and proportions of 40 bacterial species by checkerboard DNA-DNA hybridization. Differences in clinical and microbiological parameters between groups and over time were evaluated using the ANOVA, ANCOVA, Chi-square and Tukey tests. Microbiological analyzes were performed using adjustments for multiple comparisons. Statistical significance was set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age;
* at least 15 teeth (excluding third molars and teeth with advanced decay indicated for extraction);
* a minimum of 6 teeth with at least one site each with probing depth (PD) and clinical attachment level (CAL) ≥5 mm;
* at least 30% of the sites with PD and CAL ≥4 mm and bleeding on probing (BOP).

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* current smoking and former smoking within the past 5 years;
* systemic diseases that could affect the progression of periodontitis (e.g. diabetes, immunological disorders, osteoporosis);
* scaling and root planing in the previous 6 months;
* antibiotic therapy in the previous 6 months;
* long-term intake of anti-inflammatory medications;
* need for antibiotic pre-medication for routine dental therapy;
* use of orthodontic appliances;
* extensive dental prosthetic rehabilitation;
* allergy to metronidazole and/or amoxicillin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-01-31 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects reaching ≤ 4 periodontal sites with probing depth (PD) ≥ 5 mm. | 12 months

SECONDARY OUTCOMES:
Number of sites with PD ≥ 5 mm. | Baseline, 3, 6 and 12 months.
Number of sites with PD ≥ 6 mm. | Baseline, 3, 6 and 12 months.
Number of sites with PD ≥ 7 mm. | Baseline, 3, 6 and 12 months.
Reduction in the number of sites with PD ≥ 5 mm. | Baseline, 3, 6 and 12 months.
Reduction in the number of sites with PD ≥ 6 mm. | Baseline, 3, 6 and 12 months.
Reduction in the number of sites with PD ≥ 7 mm. | Baseline, 3, 6 and 12 months.
Mean PD changes in sites with initial PD between 4-6 mm | Baseline - 12 months.
Mean PD changes in sites with initial PD ≥ 7 mm. | Baseline - 12 months.
Mean CAL changes in sites with initial CAL between 4-6 mm , | Baseline - 12 months.
Mean CAL changes in sites with initial CAL ≥ 7 mm. | Baseline - 12 months.
Full-mouth PD. | Baseline, 3, 6 and 12 months.
Full-mouth clinical attachment level. | Baseline, 3, 6 and 12 months.
Percentage of sites with bleeding on probing. | Baseline, 3, 6 and 12 months.
Percentage of sites with plaque accumulation. | Baseline, 3, 6 and 12 months.
Percentage of sites with marginal bleeding. | Baseline, 3, 6 and 12 months.
Occurrence of headache obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of vomiting obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of diarrhea obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of metallic taste obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of nausea obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of irritability obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Proportions of periodontal pathogenic bacterial species. | Baseline, 3, 6 and 12 months.
Counts of periodontal pathogenic bacterial species. | Baseline, 3, 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Faveri, Professor, Study Chair — University of Guarulhos
Locations (1):
- University of Guarulhos, Guarulhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S162-S170. doi: 10.1111/jcpe.12946. PMID 29926490
- [Background] Feres M, Retamal-Valdes B, Faveri M, Duarte P, Shibli J, Soares GMS, Miranda T, Teles F, Goodson M, Hasturk H, Van Dyke T, Ehmke B, Eickholz P, Schlagenhauf U, Meyle J, Koch R, Kocher T, Hoffmann T, Kim TS, Kaner D, Figueiredo LC, Doyle H. Proposal of a Clinical Endpoint for Periodontal Trials: The Treat-to-Target Approach. J Int Acad Periodontol. 2020 Apr 1;22(2):41-53. PMID 32224549
- [Result] Feres M, Figueiredo LC, Soares GM, Faveri M. Systemic antibiotics in the treatment of periodontitis. Periodontol 2000. 2015 Feb;67(1):131-86. doi: 10.1111/prd.12075. PMID 25494600
- [Result] Feres M, Soares GM, Mendes JA, Silva MP, Faveri M, Teles R, Socransky SS, Figueiredo LC. Metronidazole alone or with amoxicillin as adjuncts to non-surgical treatment of chronic periodontitis: a 1-year double-blinded, placebo-controlled, randomized clinical trial. J Clin Periodontol. 2012 Dec;39(12):1149-58. doi: 10.1111/jcpe.12004. Epub 2012 Sep 27. PMID 23016867
- [Result] Soares GM, Mendes JA, Silva MP, Faveri M, Teles R, Socransky SS, Wang X, Figueiredo LC, Feres M. Metronidazole alone or with amoxicillin as adjuncts to non-surgical treatment of chronic periodontitis: a secondary analysis of microbiological results from a randomized clinical trial. J Clin Periodontol. 2014 Apr;41(4):366-76. doi: 10.1111/jcpe.12217. PMID 24834504
- [Result] Faveri M, Figueiredo LC, Feres M. Treatment of chronic periodontitis may be improved by the adjunctive use of systemic metronidazole. J Evid Based Dent Pract. 2014 Jun;14(2):70-2. doi: 10.1016/j.jebdp.2014.04.025. Epub 2014 Apr 12. No abstract available. PMID 24913531
- [Result] Feres M, Faveri M, Figueiredo LC, Teles R, Flemmig T, Williams R, Lang NP. Group B. Initiator paper. Non-surgical periodontal therapy: mechanical debridement, antimicrobial agents and other modalities. J Int Acad Periodontol. 2015 Jan;17(1 Suppl):21-30. No abstract available. PMID 25764587
- [Result] Borges I, Faveri M, Figueiredo LC, Duarte PM, Retamal-Valdes B, Montenegro SCL, Feres M. Different antibiotic protocols in the treatment of severe chronic periodontitis: A 1-year randomized trial. J Clin Periodontol. 2017 Aug;44(8):822-832. doi: 10.1111/jcpe.12721. Epub 2017 Jul 26. PMID 28303587
- [Result] Teughels W, Feres M, Oud V, Martin C, Matesanz P, Herrera D. Adjunctive effect of systemic antimicrobials in periodontitis therapy: A systematic review and meta-analysis. J Clin Periodontol. 2020 Jul;47 Suppl 22:257-281. doi: 10.1111/jcpe.13264. PMID 31994207
- [Result] Feres M, Retamal-Valdes B, Fermiano D, Faveri M, Figueiredo LC, Mayer MPA, Lee JJ, Bittinger K, Teles F. Microbiome changes in young periodontitis patients treated with adjunctive metronidazole and amoxicillin. J Periodontol. 2021 Apr;92(4):467-478. doi: 10.1002/JPER.20-0128. Epub 2020 Oct 12. PMID 32844406